CLINICAL TRIAL: NCT00002955
Title: Modulation of 5-Fluorouracil With Trimetrexate and Leucovorin in Advanced Pancreatic Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Cancer of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065428 (3P-95-1); LAC-USC-3P951; NCI-G97-1173
Record Dates: First submitted 1999-11-01; First posted 2004-08-12 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Pancreatic Cancer
Keywords: stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Leucovorin; trimetrexate glucuronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Drug: trimetrexate glucuronate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients with advanced cancer of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate tumor response to a trimetrexate, fluorouracil and leucovorin regimen in patients with advanced pancreatic carcinoma. II. Evaluate the toxicities associated with this regimen in patients with metastatic carcinoma of the pancreas.

OUTLINE: The treatment plan consists of an IV infusion of trimetrexate, followed 24 hours later by IV infusions of leucovorin and fluorouracil. After another 24 hours oral leucovorin will be given every 6 hours for 7 doses. A treatment cycle consists of the regimen repeated weekly for 6 weeks followed by 2 weeks of rest. Treatment cycles will be repeated until disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: If 3 or more complete or partial responses are observed in the first 22 patients, an additional 11 patients may be accrued for a maximum of 33.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced pancreatic cancer with metastatic disease Bidimensionally measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Platelet count at least 100,000/mm3 Absolute granulocyte count at least 1,500/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT, SGPT and alkaline phosphatase less than 3 times upper limit of normal Serum albumin at least 3.0 g/dL Renal: Serum creatinine no greater than 1.5 mg/dL Other: Not eligible for higher priority protocol No prior malignancy within 5 years except adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective birth control No underlying medical condition precluding treatment

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior or concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy No prior radiotherapy to only site(s) of measurable disease Fully recovered from therapy Surgery: Fully recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1995-08; Primary Completion 2000-05 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Study Chair — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Result] Garcia AA, Leichman L, Baranda J, et al.: Phase II study of trimetrexate (neutrexin), 5-fluorouracil and leucovorin (NFL) in advacne pancreatic. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A971, 253a, 1999.